CLINICAL TRIAL: NCT00354042
Title: A Randomised, Double-Blind, Placebo-Controlled, Dose Ascending, 4 Period Crossover Study to Examine the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Repeat Inhaled Doses of GW597901X in Asthmatic Subjects
Brief Title: Effects Of Repeat Inhaled Doses Of GW597901X On Patient Safety And Lung Function In Asthmatic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2A100517
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Asthma
Keywords: GW597901X; Asthma; Crossover; dose ascending; repeat dose; inhaled
MeSH Terms: conditions — Asthma; Respiratory Aspiration

INTERVENTIONS:
Drug: GW597901X

SUMMARY:
This study is designed to look at the safety aspects and effects of repeat inhaled doses of GW597901X in asthmatics to develop this drug for its use in asthma and Chronic Obstructive Pulmonary Disease(COPD).

ELIGIBILITY:
Inclusion criteria:

* Subjects with mild to moderate stable asthma but no other lung problems.
* Male subjects or female subjects who are not able to get pregnant (e.g. post-menopausal or surgically sterile).
* Non-Smokers.
* Subjects who show a measurable improvement in the function of their lungs after a single dose of salbutamol.

Exclusion criteria:

* Any significant illness.
* Subjects with heart problems.
* Subjects who have a cold or chest infection 2-4 weeks prior to the study or have life-threatening asthma.
* Subjects who take medication for their asthma, or other conditions, not compatible with this study.
* Subjects who are over sensitive to salbutamol or to ipratropium.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-08

PRIMARY OUTCOMES:
Safety Tolerability including blood test results, effects on the heart, pulse rate and blood pressure, and any side effects.

SECONDARY OUTCOMES:
Effects on the lungs at 12 and 24 hours Effects on the heart, blood pressure and heart rate at 8 hours Effects on blood tests over 4 hours and 8 hours Reduction of rescue medication.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, MSc, FPPM, Study Director — GlaxoSmithKline